CLINICAL TRIAL: NCT05179109
Title: Robotic Versus Laparoscopic Surgery for Severe Deep Endometriosis: a Prospective, Randomized, Controlled Trial
Brief Title: Robotic Versus Laparoscopic Surgery for Deep Endometriosis
Acronym: ROBEndo
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Responsible Party: Principal Investigator, Sari Koivurova, Assistant Chief of Gynecology, University of Oulu
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ROBtrial1
Record Dates: First submitted 2021-12-07; First posted 2022-01-05 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Endometriosis; Deep Endometriosis; Surgery
Keywords: Endometriosis surgery; Deep endometriosis surgery; Robotic surgery
MeSH Terms: conditions — Endometriosis | interventions — Minimally Invasive Surgical Procedures

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, controlled clinical trial with an allocation ratio of 1:1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robot-assisted laparoscopy (Experimental): Surgery for deep endometriosis using robot-assisted laparoscopy.
  Interventions: Procedure: Minimally invasive surgery
- Conventional laparoscopy (Active Comparator): Surgery for deep endometriosis using conventional laparoscopy.
  Interventions: Procedure: Minimally invasive surgery

INTERVENTIONS:
Procedure: Minimally invasive surgery — Minimally invasive surgery for severe deep endometriosis

SUMMARY:
The objective of this study is to examine whether robot-assisted laparoscopy is superior compared to conventional laparoscopy as regards to patient outcome.

DETAILED DESCRIPTION:
The objective of this prospective, randomized trial is to examine whether robot-assisted laparoscopy is superior compared to conventional laparoscopy as regards to patient outcome at 6, 12 and 24 months postoperatively, measured by questionnaires concerning the pain symptoms and disease-related quality-of life.

ELIGIBILITY:
Inclusion Criteria:

* ASA (American Society of Anesthesiologists physical status classification) 1-3
* Diagnosed deep endometriosis (MRI)
* Patient has symptoms
* Operative treatment is indicated
* Patient is able to give informed consent

Exclusion Criteria:

* ASA > 3
* Recurring rectosigmoid endometriosis

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-10-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
NRS (Numeric rating scale) Score for pain | Immediately postoperatively (24 hours) and 6, 12 and 24 months postoperatively
  The surgical outcome as regards to pain symptoms (NRS questionnaire), absolute scores and change from baseline for both study groups.

SECONDARY OUTCOMES:
Intraoperative measures | Up to 300 minutes (intraoperative)
  Operation time (minutes), blood loss (ml), complications (classified according to Clavien-Dindo) for both study groups.
Factors concerning ERAS (Enhanced recovery after surgery) | Up to 7 days (Hospital stay)
  Nausea (yes/no), vomiting (yes/no), peroral intake (minutes from surgery), mobilization (minutes from surgery), bowel movement (minutes from surgery), time of discharge (hours after surgery), complications (classified according to Clavien-Dindo) for both study groups.
Cost | Primary hospital stay and 24 months, for both study groups.
  Cost, euros.
Complications | 30 days
  Complications (classified according to Clavien-Dindo), readmissions to hospital.
Endometriosis-related quality-of-life | 6, 12 and 24 months
  Quality-of-life questionnaire (EHP-30, Endometriosis-related health profile) described as absolute scores and change from the baseline. Scale 0-100. Score 0 equals the best outcome and score 100 equals the worst outcome.
General 15 dimensional health-related quality-of-life questionnaire | 6, 12 and 24 months
  Quality-of-life questionnaire (15D, general quality-of-life questionnaire) described as absolute scores and change from baseline for both study groups. Scale 0-1. Score 0 equals the worst outcome and score 1 equals the best outcome.
Sexual quality-of-life questionnaire | 6, 12 and 24 months
  Quality-of-life (FSFI, female sexual function index) described as absolute scores and change from baseline for both study groups. Scale 2,0-36,0. Score 2,0 equals the worst outcome and score 36,0 equals the best outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Sari Koivurova, MD, PhD, Principal Investigator — Oulu University Hospital, Department of Obstetrics and Gynecology
Locations (1):
- Northern Ostrobothnia Hospital District, Oulu, Finland

REFERENCES:
- [Derived] Terho AM, Makela-Kaikkonen J, Ohtonen P, Uimari O, Puhto T, Rautio T, Koivurova S. Robotic versus laparoscopic surgery for severe deep endometriosis: protocol for a randomised controlled trial (ROBEndo trial). BMJ Open. 2022 Jul 18;12(7):e063572. doi: 10.1136/bmjopen-2022-063572. PMID 35851028